CLINICAL TRIAL: NCT06387511
Title: NutriVax-Measles: Increasing Measles Vaccination Coverage Through Supplementation With an SQ-LNS Incentive in Children Aged 6-23 Months, a Pragmatic Parallel Cluster-randomized Controlled Trial in Yobe State, Northern Nigeria
Brief Title: Increasing Measles Vaccination Coverage Through Supplementation With an SQ-LNS Incentive in Children Aged 6-23 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for International Medical Action (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Programme PAC-CI, Site ANRS-MIE de Côte d'Ivoire (Other); Yobe State Primary Health Care Board, Nigeria (Unknown); Eleanor Crook Foundation, ECF (Unknown); Gavi, The Vaccine Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NutriVax-Measles
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Immunization Coverage; Vaccination; Nutrition
Keywords: Vaccination coverage; Incentives; Small quantity of Lipid Based Nutrients (SQ-LNS); Measles; Cost-effectiveness; Acceptability; Child; Africa; Nigeria; Malnutrition, prevention
MeSH Terms: conditions — Measles; Malnutrition

STUDY DESIGN:
Intervention Model Description: A two arms superiority opened pragmatic parallel cluster-randomized controlled trial with baseline measure
Masking Description: No possible to mask intervention due to the specifity of the intervention tested
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Expanded program on immunization (Active Comparator): The standard Expanded Program on Immunization (EPI) in children aged 6-23 months delivered according to the Ministry of Health's routine plans in the community and at health centres and health posts.
  Interventions: Behavioral: Sensitization on vaccination and on Infant and Young Child Feeding (IYCF) practices
- NutriVax (Experimental): The NutriVax strategy combines the EPI in children aged 6-23 months according to the Ministry of Health's routine plans in the community and at health centres and health posts associated with SQ-LNS mass supplementation integrated into pre-existing services delivered at health centres for children 6-23 months of age.
  Interventions: Dietary Supplement: Small-quantity lipid-based nutrition supplements (SQ-LNS) NutriVax; Behavioral: Sensitization on vaccination and on Infant and Young Child Feeding (IYCF) practices

INTERVENTIONS:
Dietary Supplement: Small-quantity lipid-based nutrition supplements (SQ-LNS) NutriVax — 1. The SQ-LNS distribution program will be implemented for 12 consecutive months in the NutriVax arm.
  2. Community mobilizers in the NutriVax arm will give information in the community about SQ-LNS and eligibility criteria for SQ-LNS distributions.
  3. All SQ-LNS distributions will take place at the primary health care center (PHCC) of each ward.
  4. Children aged 6-22m, residing in settlements of the catchment area of the NutriVax arm are eligible for a monthly ration of SQ-LNS (28 sachets per month) following a check and update of his or her vaccine status at PHCC; unless there are serious issues related to access to PHCC, in which cases ration sizes may be revised upwards to three months' worth.
  5. All children will exit the SQ-LNS distribution program when they are 23 months of age OR after receiving a maximum of 12 consecutive monthly rations, whichever comes first.
  6. The total amount of SQ-LNS a child receives will depend on when they enroll in the SQ-LNS distribution program.
  Arms: NutriVax
Behavioral: Sensitization on vaccination and on Infant and Young Child Feeding (IYCF) practices — 1. Parents or guardian of children will be encouraged/sensitised to attend their scheduled preventive visits to receive other essential paediatric services;
  2. Sensitization on vaccination and recommended Infant and Young Child Feeding (IYCF) practices including the need to consume a diverse nutritious diet and support for continued breastfeeding will be conducted according to the Ministry of Health's routine plans in the community and at primary health care centres;
  3. Community mobilizers will promote the importance of vaccinations according to the Expanded Program on Immunization (EPI) as well as IYCF good practices messages.

SUMMARY:
Provision of SQ-LNS also holds promise in incentivizing vaccination as well as other health services.

The investigators will estimate 1) the effectiveness of a SQ-LNS mass supplementation program added to routine immunization program compared to routine immunization program alone in terms of measles vaccine coverage, after 12 months of program implementation, 1) in children aged 12-23 months in the end line cross-sectional household survey, 2) in children aged 6-12 months at inclusion, in a longitudinal 12 months follow-up survey.

Secondary objectives are to assess the barriers and facilitators from the perspectives of parents/legal guardian of children, health care providers and community health workers and to assess the cost-efficiency of the

This study will be implemented in 20 wards covering the Karasuwa and Nguru Local Government Areas (LGAs) in Yobe state, Northeast Nigeria.

This is a pragmatic parallel cluster randomized trial (PCT) with baseline measure with different populations and data collection modes: 1) baseline and end line cross-sectional household surveys of children aged 12-23 months, 2) a longitudinal follow-up survey (LS) of children aged 6-12 months at inclusion, 3) a qualitative feasibility and acceptability survey of parents of children aged 6-23 months, of health providers, of community health workers and community representatives and 4) a cost survey of parents/legal guardian of children from the longitudinal follow-up cohort, and 5) a health facility cost survey of a randomized subsample of health facilities.

Clusters will be randomly allocated at a ratio of 1:1 either to the standard arm or to the NutriVax arm:

* The standard Expanded Program on Immunization (EPI) in children aged 6-23 months delivered according to the Ministry of Health's routine plans in the community and at health centres and health posts, named the standard EPI arm;
* The NutriVax program combining the EPI in children aged 6-23 months according to the Ministry of Health's routine plans in the community and at health centres (i.e. PHCCs) and health posts associated with SQ-LNS mass supplementation integrated into pre-existing services delivered at health centres (i.e. PHCCs) for children 6-23 months of age, named the NutriVax arm.

DETAILED DESCRIPTION:
Background/ Rational

Every year, hundreds of thousands of children are treated for severe wasting while experiencing repeated and prolonged outbreaks of vaccine-preventable illnesses, most notably measles. At least 20 million children annually still do not receive immunizations. Northeast Nigeria is at the epicentre of this dynamic, recording some of the worst malnutrition indicators and lowest vaccination coverage rates in the world.

Small-quantity lipid-based nutrient supplements (SQ-LNS) are a class of ready-to-use food supplements which are highly nutrient-dense and fortified designed for preventing malnutrition and improving child survival, growth, and development. A recent meta-analysis on SQ-LNS reveals that feeding a child just one sachet of SQ-LNS a day for a year can reduce their risk of mortality by 27%, and reduce cases of severe wasting by 31% and severe stunting by 17%. The overall strength of evidence on SQ-LNS benefits led the authors of a 2021 Lancet review to call scaling-up SQ-LNS a priority action.

Provision of SQ-LNS also holds promise in incentivizing vaccination as well as other health services.

Primary objective

To estimate the effectiveness of a SQ-LNS mass supplementation program added to routine immunization program compared to routine immunization program alone in terms of measles vaccine coverage, after 12 months of program implementation, in children aged 12-23 months in the end line cross-sectional household survey.

Main secondary objective

To estimate the effectiveness of a SQ-LNS mass supplementation program added to routine immunization program compared to routine immunization program alone in terms of measles vaccine coverage, after 12 months of program implementation, in children aged 6-12 months at inclusion in the longitudinal 12 months follow-up survey.

Secondary objectives

* To estimate the effectiveness of a SQ-LNS mass supplementation program added to routine immunization program compared to routine immunization program alone in children aged 6-23 months, after 12 months of program implementation, in terms of 1) all other infant vaccines' uptake, 2) timeliness of age-eligible vaccinations; 3) anthropometric status, 4) uptake of paediatric curative and preventive health consultations and activities.
* To assess the barriers and facilitators to SQ-LNS mass supplementation implemented as part of a routine immunization program in health facilities, from the perspectives of parents/legal guardian of children aged 6-23 months, health care providers and community health workers.
* To assess the cost-efficiency of a SQ-LNS mass supplementation program compared to routine immunization program in terms of cost per child supplemented and vaccinated.

Study sites : 20 wards covering the Karasuwa and Nguru Local Government Areas (LGAs) in Yobe state, Northeast Nigeria

Study design

A pragmatic parallel cluster randomized trial (PCT) with baseline measure with different populations and data collection modes: 1) baseline and end line cross-sectional household surveys of children aged 12-23 months, 2) a longitudinal follow-up survey (LS) of children aged 6-12 months at inclusion, 3) a qualitative feasibility and acceptability survey of parents of children aged 6-23 months, of health providers, of community health workers and community representatives and 4) a cost survey of parents/legal guardian of children from the longitudinal follow-up cohort, and 5) a health facility cost survey of a randomized subsample of health facilities.

Interventions compared

1. The standard Expanded Program on Immunization (EPI) in children aged 6-23 months delivered according to the Ministry of Health's routine plans in the community and at health centres and health posts, named the standard EPI arm.
2. The NutriVax program combining the EPI in children aged 6-23 months according to the Ministry of Health's routine plans in the community and at health centres (i.e. PHCCs) and health posts associated with SQ-LNS mass supplementation integrated into pre-existing services delivered at health centres (i.e. PHCCs) for children 6-23 months of age, named the NutriVax arm.

The unit of randomization (cluster) will be the ward and its catchment area. Clusters will be randomly allocated at a ratio of 1:1 either to the standard EPI arm or to the NutriVax arm.

Statistical analyses

Differences in measles vaccine coverage (dose 1) between control and intervention arms at end line will be assessed using multilevel regression models.

The study will be conducted in compliance with the protocol, the Declaration of Helsinki, the GCP guidelines and the Nigerian National Code for Health Research Ethics

Timeline : 2 years (December 2023-December 2025)

ELIGIBILITY:
* Baseline and endline cross-sectional household surveys Inclusion criteria

  * Aged 12-23 months;
  * With oral informed consent of parent or legal guardian;
  * Residing in the catchment settlements of wards included in the study. Exclusion criteria
  * Included in the longitudinal follow-up.
* Longitudinal follow-up survey Inclusion criteria

  * Aged 6-12 months;
  * With written informed consent of parent or legal guardian;
  * Residing in the catchment settlements of wards included in the study. Exclusion criteria
  * Acute malnutrition criteria as per the WHO definition (i.e. MUAC< 125 or WHZ < -2 or nutritional edema);
  * - Known medical complication that requires referral for hospitalization;
  * Known allergies to SQ-LNS or SQ-LNS contraindication;
  * Any other condition interfering with protocol adherence or the ability to give informed consent, in the judgment of the Field Investigator Sampling for HHS and LS will be carried out in three stages in each LGA using probability proportional to size (PPS).
* Qualitative feasibility and acceptability survey Inclusion

  * Parent or legal guardian of a child aged 6-23 months and residing in the catchment settlements of wards included in the study, or Health worker of the ministry of health involved in the study,or Community representative or Community health workers;
  * With written informed consent.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3814 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Measles vaccine coverage in children aged 12-23 months | Measured after one year after of intervention implementation.
  The proportion of children aged 12-23 months in the endline survey who have received at least one dose of measles vaccine, as reported on their vaccination card.
Measles vaccine coverage in children 6-12 months at inclusion | Measured after one year after of intervention implementation.
  The proportion of children aged 6-12 months at inclusion in the longitudinal follow-up survey, who have received at least one additional dose of measles vaccine, as reported on their vaccination card, administered between inclusion and the end of follow-up.

SECONDARY OUTCOMES:
Measles vaccine coverage: at least one dose | Measured after one year after of intervention implementation.
  The proportion of children with at least one measles vaccine as reported on a vaccination card or by recall.
Measles vaccine coverage : two doses | Measured after one year after of intervention implementation.
  The proportion of children with a measles 2 vaccine as reported on a vaccination card or by recall
Timeliness of measles 1 vaccination | Measured after one year after of intervention implementation.
  Proportion of children with Measles 1 vaccine received within 30 days of turning 9 months by card
Other infant vaccines coverage | Measured after one year after of intervention implementation.
  Proportion of children with Pentavalent 1 and 3, yellow fever, meningitis vaccine as reported on a vaccination card or by recall
Zero-dose | Measured after one year after of intervention implementation.
  Proportion of children with No measles + pentavalent + yellow fever + meningitis vaccines reported on a vaccination card or by recall.
Fully immunization | Measured after one year after of intervention implementation.
  Proportion of children who had received all childhood vaccinations recommended by the Nigeria MOH.
Acceptability | Measured after 2 months and one year after of intervention implementation.
  Barriers and facilitators to access health care centres and receive SQ-LNS mass supplementation implemented as a routine preventive program nested in health facilities activities
Cost-efficiency | Measured after one year after of intervention implementation.
  • Cost per child vaccinated and supplemented compared to cost per child vaccinated only, using a facility and caregiver perspectiveto identify all provider and caregiver costs associated with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Becquet, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- All Primary Health Care Centers of Nguru and Karasuwa LGAs, Damaturu, Yobe State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Possible data sharing agreement, possible one year after publication of the main results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before (protocol, ICF) and during data collection (SAP)
Access Criteria: Protocol, ICF and SAP on clinicaltrials.gov

REFERENCES:
- [Derived] Cazes C, Goni BW, Muhammad NS, Gabillard D, Balonda PK, Feuzeu L, Atanga I, Yapi B, Habiyambere GG, Danho S, Balestre E, Adams KP, Plazy M, Phelan KPQ, Becquet R. Increasing measles vaccination coverage through supplementation with an SQ-LNS incentive in children aged 6 to 23 months: study protocol of NutriVax-Measles, a superiority pragmatic parallel cluster-randomized controlled trial in Yobe State, Northern Nigeria. Trials. 2025 Nov 19;26(1):525. doi: 10.1186/s13063-025-09243-5. PMID 41257898
- See also: Resource: A Review & Proposed Learning Agenda on Immunization Nutrition Integration — https://eleanorcrookfoundation.org/the-latest/resources/a-literature-review-on-immunization

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT06387511/SAP_000.pdf